CLINICAL TRIAL: NCT01238055
Title: Randomized Phase II Trial of Sunitinib and Docetaxel in Advanced Gastric Cancer Patients Who Had Prior Chemotherapy With Fluoropyrimidine and Platinum
Brief Title: Sunitinib + Docetaxel as Second-line Treatment in Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-09-031
Record Dates: First submitted 2010-01-07; First posted 2010-11-10 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2012-01

CONDITIONS: Advanced Gastric Cancer
Keywords: advanced gastric cancer; sunitinib; docetaxel; fluoropyrimidine platinum based chemotherapy
MeSH Terms: interventions — Docetaxel; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel + Sunitinib (Experimental): Docetaxel and Sunitinib
  Interventions: Drug: Docetaxel + Sunitinib
- Docetaxel (Active Comparator): Docetaxel only
  Interventions: Drug: Docetaxel only

INTERVENTIONS:
Drug: Docetaxel + Sunitinib — Docetaxel 60 mg/m2 iv, every 3 weeks
  Sunitinib 37.5 mg qd daily, every 3 weeks
  Arms: Docetaxel + Sunitinib
Drug: Docetaxel only — Docetaxel 60 mg/m2 iv
  Arms: Docetaxel

SUMMARY:
The purpose of this study is to determine whether Sunitinib and Docetaxel is effective in the treatment of advanced gastric cancer patients who had prior chemotherapy with fluoropyrimidine and platinum.

DETAILED DESCRIPTION:
This is a randomized phase II trial of Sunitinib and Docetaxel in advanced gastric cancer patients who had prior chemotherapy with Fluoropyrimidine and Platinum.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or cytologically confirmed diagnosis of gastric adenocarcinoma or gastroesophageal junction adenoca (i.e. an adenocarcinoma with > 50% extension in the stomach)
2. patients must present with stage IV disease not amenable to surgery, radiation or combined modality therapy with curative intent. Patients previously undergoing local treatment (surgery and/or radiation) must have subsequently progressed or recurred
3. prior chemotherapy wit fluoropyrimidine and platinum
4. measurable or evaluable disease according to RECIST
5. age, 18 years or older
6. ECOG performance status 0 - 2
7. adequate organ function as defined by the following criteria absolute neutrophil count (ANC) ≥ 1,500/ul platelets ≥ 100,000/ul AST/ALT ≤ 2.5 x ULN, ≤ 5.0 x ULN if liver involvement Total serum bilirubin ≤ 2.0 mg/dL
8. life expectancy of ≥ 3 months
9. signed written informed consent

Exclusion Criteria:

1. more than one prior chemotherapy for metastatic disease
2. severe co-morbid illness and/or active infections
3. NCI CTCAE Grade 3 hemorrhage from any cause < 4 weeks before enrollment
4. preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart
5. pregnant or lactating women
6. active CNS metastases not controllable with radiotherapy or corticosteroids
7. active and uncontrollable bleeding from gastrointestinal tract
8. known history of hypersensitivity to study drugs
9. prior treatment with sunitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-11; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
time to progression | every 6 weeks

SECONDARY OUTCOMES:
Response rate | 12 months
Overall survival | 12 months
Progression free survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea